CLINICAL TRIAL: NCT02579954
Title: Cardiac Function and Exercise Capacity in Pulmonary Arterial Hypertension
Acronym: FONCE-HTAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1308156; 2014-A00169-38 (Other: ANSM)
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- intervention (Experimental): Rehabilitation
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation
  Other Names: Supervised rehabilitation
  Arms: intervention

SUMMARY:
Pulmonary Arterial Hypertension is characterized by a progressive increase in pulmonary vascular resistance inducing shortness of breath and exercise intolerance. We aim to correlate cardiac function (evaluated at rest by right heart catheterism and RMN) to exercise capacity (evaluated by endurance time at 75% of maximal workout), in prevalent patients with pulmonary arterial hypertension, and their evolution at three and twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients with Pulmonary Arterial Hypertension (idiopathic, heritable or due to anorexigens),
* Prevalent cases of pulmonary artery hypertension (≥ 6 months) confirmed by right heart catheterism,
* Stable for at least 3 months,
* Written consent.

Exclusion Criteria:

* Patients unable to proceed with six-minute walk test or CPET, or with contra-indication to exercise evaluation (syncope, low cardiac index, etc).
* Exercise induced abnormality (evaluated during the initial CPET) precluding to further evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Endurance time at 75% of the maximal workout (determinated during a cardiopulmonary exercise testing - CPET), | 12 months after the inclusion

SECONDARY OUTCOMES:
Right ventricular ejection fraction evaluated by RMN | at 3 and 12 months
Pulmonary haemodynamics : measurements at right heart catheterism | at 3 and 12 months
  cardiac index (L/min/m²)
Pulmonary haemodynamics : measurements at right heart catheterism | at 3 and 12 months
  pressure in the right atrium (mmHg)
Pulmonary haemodynamics : measurements at right heart catheterism | at 3 and 12 months
  pulmonary resistance (uw)
Pulmonary haemodynamics : measurements at right heart catheterism | at 3 and 12 months
  mean pulmonary arterial pressure (mmHg)
Functional class (NYHA classification) | at 3 and 12 months
6 minutes walking distance (m) | at 3 and 12 months
Functional exercise capacity (oxygen consumption measurement during test) | at 3 and 12 months
Quality of life (SF-36 scale) | at 3 and 12 months
Time to clinical worsening (months) | at 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BERTOLETTI, MD PhD, Principal Investigator — CHU de Saint Etienne
Locations (10):
- France (10):
  - CHU de Besançon, Besançon
  - CHU de Brest, Brest
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Hôpital Sud de Grenoble, Échirolles
  - Hôpital Nord de Grenoble, Grenoble
  - HCL - Hôpital Louis Pradel, Lyon
  - CHU de Montpellier, Montpellier
  - APHP - Hôpital Bicêtre, Paris
  - Chu de Saint Etienne, Saint-Etienne
  - CHRU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No